CLINICAL TRIAL: NCT05380817
Title: Stanford Kids Continuous Advanced Metabolic Profiling (CAMP) Study
Brief Title: Stanford Kids CAMP Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Karl Sylvester, Associate Dean Maternal Child Health - Research, Professor of Surgery, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 65748
Record Dates: First submitted 2022-05-09; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Pre-diabetes; Obesity; Type-2 Diabetes Mellitus
MeSH Terms: conditions — Glucose Intolerance; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BAWSI Group (Other): By partnering with a community sports club (BAWSI), will the partnership recruitment model be effective in enrolling minority children.
  Interventions: Other: Remote Monitoring Program
- YMCA of Silicon Valley Group (Other): By partnering with a community organization (YMCA of Silicon Valley), will the partnership recruitment model be effective in enrolling minority children.
  Interventions: Other: Remote Monitoring Program

INTERVENTIONS:
Other: Remote Monitoring Program — Participants receive remote monitoring while engaging in a theory-based, multi-component, multi-level, multi-setting (MMM) community team sports program designed specifically for children

SUMMARY:
The Stanford Kids CAMP study aims to evaluate the feasibility of enrolling minority participants in school age children (5-13 years old) in a community summer camp setting along with the efficiency by which each participant's biologic specimens are collected. Using remote monitoring technologies and through partnering with community-based organizations, the investigators hypothesize that an increase in underrepresented minority participation in a clinical trial that is greater than the national average is possible.

DETAILED DESCRIPTION:
The proposed study is an outpatient prospective, open-label clinical trial comparing 2 groups: Group 1 (aka BAWSI Camp): the Dexcom G6 Pro Continuous Glucose Monitor and the accelerometer and mobile connected device, Group 2 (aka YMCA of Silicon Valley Camp): the Abbott FreeStyle Libre 2 Continuous Glucose Monitor and the accelerometer and mobile connected device. Eligible subjects will be enrolled to each cohort based on their participation in the specific YMCA camp site.

The investigators will study up to 100 minority school-age children (5 - 13 years old) in the San Francisco Bay Area a 5-day summer camp. The study will be split in 2 sequential phases: (A) the BAWSI camp, (B) the YMCA of Silicon Valley camp, following a repeated measures design with the 5-day camp being followed by 5 - 9 days at home, under parental supervision. Study participants will be divided in two equal groups at each site with each wearing the specific manufacturers continuous glucose monitoring device.

ELIGIBILITY:
Inclusion Criteria:

* 5-13 years of age.
* Avoidance of acetaminophen-containing medications (i.e. Tylenol) while wearing the continuous glucose monitor.
* Willingness to wear a continuous glucose sensor and physiological monitor for the duration of the study.
* A parent/caregiver is available for system training and will commit to be the main responsible person for the use of the monitoring system at home.

Exclusion Criteria:

* Have a condition limiting their participation in the interventions (e.g., unable to participate in routine physical education classes at school, requiring oxygen supplementation for exertion, developmental or physical disability preventing participation in interventions, children or parents/guardians who cannot medically participate in mild dietary restrictions and/or increased physical activity for any reason).
* Have a condition limiting participation in the assessments (child or primary caregiver not able to read surveys in English or Spanish, child two or more grade levels delayed in school for reading and writing in her native language).
* Are unable to read, understand or complete informed consent in English or Spanish.
* Are deemed to have another characteristic that makes them unsuitable for participation in the study in the judgment of the Principal Investigators.

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of underrepresented minority participants enrolled | Baseline (prior to arrival at camp)
  Percentage of underrepresented minority participants enrolled compared to the U.S. national average.

SECONDARY OUTCOMES:
Duration of initial participant screening | Visit 1 (day 1, up to 60 minutes for screening)
  Average duration of time to screen enrolled subjects on Day 1 of summer camp.
Report of issues and concerns during at-home monitoring period | Visit 4, Visit 6 (days 6 and 14, up to 30 minutes to complete survey)
  # of telephone reported incidents and questions during at-home monitoring period.
Physical activity measured by accelerometry | Baseline through Visit 6 (days 1 through 14)
  Garmin Vivofit 4 total and after camp physical activity and sedentary behavior
Participant perceived use of study technology | Visit 6 (day 14, up to 15 minutes to complete survey)
  Percentage of survey responses
At-home urine specimen collection | Visit 1, Visit 3 (collected on days 1 and 5)
  Percentage of enrolled participants who complete at home urine sample collection and bring the sample with them to camp.
Continuous patient monitoring performance | Baseline through Visit 6 (days 1 though 14)
  Percentage of total study time children were monitored using glucose and accelerometry devices
Number of patient reported device related issues | Visit 1, Visit 2, Visit 3 (days 1 though 5)
  This measure is intended to evaluate study device performance during summer camp

CONTACTS AND LOCATIONS:
Overall Officials: Karl Sylvester, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators can request the limited public access data set from the Stanford Metabolic Health Center's Data Coordinating Center
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data is currently unavailable.